CLINICAL TRIAL: NCT04182984
Title: TheRapeutic Effect of Different immunosuppressAnts on Non-Thymoma Ocular Myasthenia Gravis: a Real-world Study
Acronym: TREAT-OMG
Status: Recruiting | Type: Observational
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Principal Investigator, Jun Guo, MD, Associate Professor, Tang-Du Hospital
Other Study IDs: 2019TDSNOMG
Record Dates: First submitted 2019-11-26; First posted 2019-12-02 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Ocular Myasthenia Gravis
Keywords: Ocular myasthenia gravis
MeSH Terms: conditions — Myasthenia Gravis | interventions — Steroids; Tacrolimus; Mycophenolic Acid; Pyridostigmine Bromide; Prednisone; Azathioprine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with autoimmune ocular MG: Newly-onset OMG patients who agreed to join the follow-up cohort
  Interventions: Drug: Symptomatic Treatment, Steroids, Immunosuppressive Agents( azathioprine, tacrolimus, Mycophenolate Mofetil)

INTERVENTIONS:
Drug: Symptomatic Treatment, Steroids, Immunosuppressive Agents( azathioprine, tacrolimus, Mycophenolate Mofetil) — Treatment regimens are determined according to the physician's judgment and preferences of the patients.
  Other Names: Pyridostigmine Bromide, Prednisone,Azathioprine, Tacrolimus, Mycophenolate Mofetil,

SUMMARY:
This study collects the clinical data of new-onset ocular myasthenia gravis (OMG) patients, assesses outcomes and adverse effects of different treatment options, and evaluate risk factors of conversion to generalized MG(GMG).

DETAILED DESCRIPTION:
This is a multicenter, observational cohort trial in the real-world clinical setting recruiting new-onset OMG patients from Neurology Departments of 7 hospitals in different regions of China. Clinical manifestations, laboratory test results, chest imaging and history of thymectomy are recorded. Treatment option are determined according to the physician's judgment and preferences of the patients. Patients are followed up prospectively on regular to assess the outcomes of treatments and monitor any side effects. Peripheral blood samples are collected annually. The investigators plan to recruit a final sample of 200 patients for analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years and<75 years;
2. Clinical Diagnosis of MG with supporting evidence:

   Patients with ocular muscle type MG who have never received treatment meet one of the diagnoses (1) and (2)-(5): (1) The patient's symptoms involve the extraocular muscles, except for drooping eyelids and diplopia, no other clinical symptoms; (2) unequivocal clinical response to pyridostigmine; (3) positive acetylcholine receptor antibody or musk antibody; (4) decrement of more than 10% in repetitive nerve stimulations study (RNS); (5) the "trembling" of the single fiber electromyography (SFEMG) is broadened with or without blockade;
3. Willingness to sample collection, imaging study and other disease-related examinations and assessments;
4. The results of pregnancy tests for female subjects with fertility during the screening period should be negative and effective contraception was used by the patient and her spouse during the study period;
5. Patients with informed consent;
6. Predicted survival time is longer than 3 years.

Exclusion Criteria:

1. History of chronic degenerative, psychiatric, or neurologic disorder other than MG that can produce weakness or fatigue;
2. Patients who may have other diseases that may lead to eyelid drooping, peripheral muscle weakness or diplopia;
3. Age ≤18 years or ≥75 years;
4. Patients who have been taking glucocorticoids or associated immunosuppressants due to other immune system diseases;
5. Patients who cannot use immunosuppressants due to other chronic diseases;
6. Patients who are unable to cooperate with follow-up and self-assessment due to severe mental illness or cognitive impairment;
7. Pregnant women, lactating women and patients with fertility plans during the trial;
8. Patients who have suffered from severe infections or malignant tumors in the last 1 month and are unable to receive immunosuppressants treatments;
9. Patients who are not willing to cooperate with repeated frequency electrical stimulation tests and chest CT examinations;
10. Patients who are not willing to participate in this study;
11. Patients who are unable to sign informed consent;
12. Predicted survival time is shorter than 3 years;
13. Patients who are not suitable to participated in the trial after researchers' assessment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly-onset ocular myasthenia gravis
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-11-04 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Conversion rate from ocular to generalized MG at the last follow-up visit. | 144 weeks
  Ocular MG patients are followed up to determine the ratio of conversion to generalized disease at the end of follow-up. The clinical records will be retrospectively analyzed to search for risk factors of progressing.
Changes in the ratio of patients who achieve the level 2 of MG Status and Treatment Intensity (MGSTI) scale or better. | Baseline, 12 weeks, 24 weeks, 36 weeks, 48 weeks, 60 weeks, 72 weeks, 96 weeks, 120 weeks, 144 weeks
  Ocular MG patients are followed up to determine the ratio of patients that achieve the status of MGSTI 2 or better at each period piont of follow-up. The clinical records will be retrospectively analyzed to search for risk factors prolonged the regimens reduction.
Changes in proportion of patients with treatment-related adverse events. | Baseline, 12 weeks, 24 weeks, 36 weeks, 48 weeks, 60 weeks, 72 weeks, 96 weeks, 120 weeks, 144 weeks
  Treatment-Related Adverse Events (AEs) are evaluated in patients receiving different treatment protocol
Changes in scores of Quantitative Myasthenia Gravis (QMG) scale and of Absolute and Relative Score of MG(ARS-MG) scales from Baseline. | 12 weeks, 24 weeks, 36 weeks, 48 weeks, 60 weeks, 72 weeks, 96 weeks, 120 weeks, 144 weeks
  The improvement of clinic status of OMG patients was assessed by investigators according to QMG and ARS-MG score. The QMG is a 13-item scale which measures ocular, bulbar, limb function and respiratory function. The total score ranges from 0 (no myasthenic findings) to 39 (maximal myasthenic deficits) obtained by summing the responses to each individual item.The ARS-MG is a 8-item scale which has a more detailed measure to assess ocular function . The total score ranges from 0 (no myasthenic findings) to 60 (maximal myasthenic deficits) obtained by summing the responses to each individual item.
Changes in scores of MG-specific Activities of Daily Living (MG-ADL) scale from Baseline. | 12 weeks, 24 weeks, 36 weeks, 48 weeks, 60 weeks, 72 weeks, 96 weeks, 120 weeks, 144 weeks
  The improvement of clinic status of OMG patients was assessed by patients themselves according to MG-ADL score. The The MG-ADL is an 8-item scale to assess symptoms of myasthenia gravis patients obtained by summing the responses to each individual item (Grades: 0,1,2,3). The score ranges from 0 to 24.

SECONDARY OUTCOMES:
Changes in titers of MG antibodies. | Baseline, 48 weeks, 96 weeks, 144 weeks
  MG antibodies are detected at enrollment and the titers of antibodies will be monitored annually.
Improvement of repeated frequency electrical stimulation tests (RNS) and single fiber electromyography (SFEMG). | 12 weeks, 24 weeks, 36 weeks, 48 weeks, 60 weeks, 72 weeks, 96 weeks, 120 weeks, 144 weeks
  RNS and SFEMG will be monitored on time to assess the clinic status.
Relapse rate during follow-up period. | Baseline, 144 weeks
  Ocular MG patients are followed up to determine the relapse rate at the end of follow-up. The clinical records will be retrospectively analyzed to search for risk factors of recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Guo, Study Chair — Tangdu Hospital, Air Force Military Medical University
Locations (1):
- Tangdu Hospotal, Xi'an, Shaanxi, China